CLINICAL TRIAL: NCT00923403
Title: Efficacy of Sterol-Fortified Low Fat Soy Beverage on Cholesterol Metabolism, Inflammation and Oxidative Status in Humans - Study II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: WhiteWave Foods, Inc. (Industry)
Responsible Party: Peter JH Jones, Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 555-210
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Hypercholesterolemia
Keywords: plant sterols; diet; soymilk; cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Comparator (Placebo Comparator): control dairy milk
  Interventions: Dietary Supplement: control dairy milk
- experimental (Experimental): plant sterol enriched soymilk
  Interventions: Dietary Supplement: plant sterol enriched soymilk

INTERVENTIONS:
Dietary Supplement: plant sterol enriched soymilk — plant sterol enriched soymilk
  Arms: experimental
Dietary Supplement: control dairy milk — control dairy milk
  Arms: Placebo Comparator

SUMMARY:
Hypercholesterolemia is a well-established risk factor for the development of atherosclerosis, a component of cardiovascular disease (CVD). The National Cholesterol Education Program advises the public to consume 2 g/day of plant sterols or stanols in addition to the Therapeutic Lifestyle Change Diet to lower elevated low-density lipoprotein (LDL) cholesterol levels. For foods to carry the FDA health claim label they must contain 0.65 g of phytosterol ester or 1.7 g of phytostanol ester per serving. The study was a controlled diet, cross-over clinical investigation using a Latin square sequence. It consisted of two 29 d phases separated by a four week wash out interval. Subjects were randomized to one of two treatment arms: 1 % dairy milk or low-fat soy beverage providing 1.95 g plant sterols/day.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, age 19-60 years old, will be screened for determination of fasting circulating LDL-cholesterol and triglyceride (TG) levels.
2. Subjects accepted into the study will have plasma LDL-C levels between 120 and 200 mg/dl, TG levels below 250 mg/dl, and a body mass index (BMI) between 22 to 32 kg/m2.
3. Subjects must also demonstrate an ability to understand dietary and exercise procedures and be judged as compliant and motivated by the investigators.
4. Subjects will be permitted to take stable doses of thyroid hormone and anti-hypertensive agents, as long as these are continued equivalently throughout the duration of study.

Exclusion Criteria:

1. History of recent (i.e. less than 3 mo) or chronic use of oral hypolipidemic therapy, including fish oils, or probucol within the last 6 months.
2. History of chronic use of alcohol (>2 drinks/d), systemic antibodies, corticosteroids, androgens, or phenytoin.
3. Myocardial infarction, coronary artery bypass, or other major surgical procedures within the last six months.
4. Recent onset of angina, congestive heart failure, inflammatory bowel disease, pancreatitis, diabetes, or significant current (ie. onset within past three months) gastrointestinal, renal, pulmonary, hepatic or biliary disease, or cancer (evidence of active lesions, chemotherapy or surgery in the past year).
5. Exercise greater than walking or running 15 miles/wk or 4,000 kcal/week.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
plasma cholesterol | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PHD, Principal Investigator — Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Rideout TC, Chan YM, Harding SV, Jones PJ. Low and moderate-fat plant sterol fortified soymilk in modulation of plasma lipids and cholesterol kinetics in subjects with normal to high cholesterol concentrations: report on two randomized crossover studies. Lipids Health Dis. 2009 Oct 20;8:45. doi: 10.1186/1476-511X-8-45. PMID 19843338